CLINICAL TRIAL: NCT07167134
Title: Evolution of Hypofractionated Stereotactic Irradiation for Radio-Resistant Brain Metastases From D1-3-5 to D1-2-3
Acronym: SISMIC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-014
Record Dates: First submitted 2025-08-21; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Brain Metastases
Keywords: hypofractionated stereotactic radiotherapy; treatment duration
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D1-3-5 radiotherapy (Active Comparator): The prescribed total dose will be 23.1 Gy delivered in 3 fractions of 7.7 Gy on days 1, 3, and 5**. The prescription will be based on 70% isodose line, resulting in a total dose of 33 Gy at the isocenter.
  Interventions: Radiation: D1-3-5 radiotherapy
- D1-2-3 radiotherapy (Experimental): The prescribed dose will be 23.1 Gy at delivered in 3 fractions of 7.7 Gy on days 1, 2, and 3*. The prescription will be based on 70% isodose line, resulting in a total dose of 33 Gy at the isocenter.
  Interventions: Radiation: D1-2-3 radiotherapy

INTERVENTIONS:
Radiation: D1-3-5 radiotherapy — 23.1 Gray (Gy) delivered in 3 fractions of 7.7 Gy at D1, D3, and D5
  Arms: D1-3-5 radiotherapy
Radiation: D1-2-3 radiotherapy — 23.1 Gray (Gy) delivered in 3 fractions of 7.7 Gy at D1, D2, and D3
  Arms: D1-2-3 radiotherapy

SUMMARY:
The goal of this prospective, multi-center, randomized double-arm clinical trial is to demonstrate a benefit in term of local control of a shorter spread of hypofractionated stereotactic radiotherapy at D1-2-3 vs D1-3-5, in the treatment of "radioresistant" Brain Metastases (BM). This trial aims to recruit patients with 1 to 5 unoperated BM originating from radioresistant primary sites. Patients will be randomly assigned to either the D1-3-5 radiotherapy arm or the D1-2-3 radiotherapy arm. Stereotactic brain irradiation will be administered at a dose of 33 Gy delivered in 3 fractions.

DETAILED DESCRIPTION:
Brain metastases (BM), originating from various primary tumors, are associated with decreased progression-free survival, overall survival, and neurological function. Stereotactic radiotherapy offers a precise and targeted approach to treat BM while minimizing cognitive side effects. Studies have shown comparable local control rates to surgery and conventional radiotherapy, but radioresistant cancers exhibit lower response rates whatever the technique of radiotherapy. The radiobiological implications of treatment duration in brain stereotactic irradiation remain understudied, resulting in a lack of available data. However, there is potential for a shorter irradiation duration to enhance tumor control without an accompanying increase in treatment-related toxicity. This study aims to demonstrate a benefit in terms of local control of a shorter spread of hypofractionated stereotactic radiotherapy at D1, D2, D3 vs D1, D3, D5, in the treatment of radioresistant brain metastases.

This prospective, multi-center, randomized, double-arm clinical trial aims to recruit patients with 1 to 5 unoperated brain metastases originating from radioresistant primary sites. Patients will be randomly assigned to either the D1,3,5 radiotherapy arm or the D1,2,3 radiotherapy arm and will be followed for 2 years. Stereotactic brain irradiation will be administered at a dose of 33 Gy delivered in 3 fractions at the isocenter.

The primary endpoint of the study is the assessment of local control at 6 months per brain metastasis. Secondary endpoints include evaluating cerebral control, overall survival, radionecrosis rate, quality of life, neurological function, and treatment-related toxicity.

A more condensed treatment approach may exploit the radiobiological properties of tumors, potentially increasing their sensitivity to radiation while minimizing the opportunity for tumor repopulation. Moreover, reducing treatment duration also has the potential to improve the patient's quality of life by minimizing fatigue towards the end of the irradiation course.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with one or more unoperated brain metastases (1-5) originating from radioresistant primary locations, including melanoma, kidney, digestive, sarcoma, and prostate *
* Karnofsky Performance Status (KPS) greater than 50% (Annex 3).
* Absence of major psychiatric conditions in the medical history that may interfere with follow-up, based on the investigator's judgement.
* Proficiency in understanding French.
* Signed informed consent.
* For the ancillary study only: Patients included in the SISMIC study at centers with adequate resources and who have agreed to participate in the optional ancillary study.

  * Note: Patients who have had one or more surgery for metastasis removal and also have unresectable metastases are eligible for inclusion. Irradiation of the operating bed will follow the same treatment regimen as existing metastases but will not be considered for the evaluation of local control.

Exclusion Criteria:

* Pregnant or breastfeeding women
* An unoperated brain metastasis whose maximum diameter is > 3.5 cm
* Patients deprived of liberty or under guardianship (including curatorship).
* Patients with a history of cerebral radiotherapy.
* Patients with known allergy to gadolinium.
* Contraindication to magnetic resonance imaging (MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Local control of brain metastases at 6 months | at 6 months
  Local control at 6 months per brain metastasis evaluated with magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Local control of brain metastases at 12, 18 and 24 months | at 12, 18 and 24 months
  Local control at 6 months per brain metastasis evaluated with magnetic resonance imaging (MRI).
Cerebral control at 12, 18 and 24 months | at 12, 18 and 24 months
  Cerebral control is defined as the assessment of the control of the entire cerebral parenchyma, including the treated site(s) evaluated with magnetic resonance imaging (MRI).
Overall survival | From the date of randomization until the date of death from any cause, loss to follow-up, or 24 months, whichever occurs first
  The time from the date of randomization to the date of death, whatever the cause. Patients alive at the time of analysis will be censored on the date of last contact.
Progression-free survival | According to local practices until the date of first documented progression or the date of death from any cause or until 24 months, whichever occurs first
  Time between the date of randomization and the date of first progression of the irradiated site (or one of the sites irradiated in the event of irradiation of several sites) or the date of death. Patients alive without progression will be censored on the last news date.
Patient Quality of life | Before radiotherapy, then at 3, 6, 12, 18 and 24 months from randomization
  Assessment of all dimensions of EORTC QLG Core Questionnaire (EORTC QLQ-C30). Difference on specific symptom scales (from 1 = " not at all " to 4 = " very much ", or from 1 = " really bad " to 7 = " excellent ")
Patient Quality of life | Before radiotherapy, then at 3, 6, 12, 18 and 24 months from randomization
  Assessment of difference on specific symptom scales of the European Organization for Research and Treatment of Cancer (EORTC) QLQ-BN20 brain tumour module questionnaire (from 1 = " not at all " to 4 = " very much).
Risk of leptomeningeal dissemination | according to local practices until death from any cause or lost to follow-up or until 24 months, whichever came first
  Local or diffuse leptomeningeal disease or positive cerebrospinal fluid examination for malignant cells based on MRI findings
Radionecrosis-free survival | according to local practices until death from any cause or lost to follow-up or until 24 months, whichever came first
  The time from the date of randomization to the date of detection of radionecrosis
Patient Safety | From the date of randomization until the date of death from any cause, loss to follow-up, or 24 months, whichever occurs first
  Incidence of treatment-related adverse events (TRAEs) graded according to CTCAE v5.0 criteria and deaths
Patient Safety according to Patient Reported Outcome | From the date of randomization until the date of death from any cause, loss to follow-up, or 24 months, whichever occurs first
  Incidence of treatment-related adverse events (TRAEs) according to patient's declaration
Cognitive decline assessment | At baseline (before radiotherapy), then at 3, 6 and 12 months from randomization
  Evaluation of neurological function by neuropsychological evaluation, centered on global deficiencies with the Montreal Cognitive Assessment (MoCA). It allows assessment of attention, concentration, executive functions, memory, language, visuoconstructive abilities, abstraction, calculation, and orientation. Maximum score = 30. A score below 26 is considered abnormal.
Cognitive decline assessment | at baseline (before radiotherapy), then at 3, 6 and 12 months from randomization
  Evaluation of neurological function by neuropsychological evaluation, centered on cognitive complaints with the Functional Assessment of Cancer Therapy - Cognitive Function (Fact-Cog) self-questionnaire. It allows assessment of Perceived Cognitive Impairments (from 0 = " never " to 4 = " several times a day "), Comments from Others (from 0 = " never " to 4 = " several times a day "), Perceived Cognitive Abilities (from 0 = " not at all " to 4 = " very much "), Impact on Quality of Life (from 0 = " not at all " to 4 = " very much ")
Cognitive decline assessment | at baseline (before radiotherapy), then at 3, 6 and 12 months from randomization
  Evaluation of neurological function by neuropsychological evaluation. Evaluations centered on information processing speed (Computerized Speed Cognitive Test - CSCT).

CONTACTS AND LOCATIONS:
Locations (1):
- ICANS, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided